CLINICAL TRIAL: NCT01108744
Title: Double Blind Study of Hypertonic Saline vs Mannitol in the Management of Increased Intracranial Pressure (ICP).
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Timeline to consent prior to intervention start was unfeasible.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Achikam Orin-Grinberg, Assistant Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009P000313
Record Dates: First submitted 2010-04-16; First posted 2010-04-22 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Elevated Intracranial Pressure
Keywords: clinical trial; mannitol; intracranial pressure (ICP); hypertonic saline; cerebral edema; traumatic brain injury (TBI)
MeSH Terms: conditions — Intracranial Hypertension; Brain Edema; Brain Injuries, Traumatic | interventions — Saline Solution, Hypertonic; Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypertonic saline (Active Comparator): 3% hypertonic saline, dosed by ideal patient weight
  Interventions: Drug: hypertonic saline
- Mannitol (Active Comparator): 20% mannitol, dosed by patient's ideal body weight
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: hypertonic saline — 3% hypertonic saline, dosed by ideal patient weight
  Arms: hypertonic saline
Drug: Mannitol — Mannitol 20% intravenous solution, dosed by patient's ideal body weight
  Other Names: Osmitrol
  Arms: Mannitol

SUMMARY:
The study goal is to compare the management of increased intra-cranial pressure (ICP) using 3% hypertonic saline vs. mannitol (given in same osmolar loads).

Primary hypothesis:

1. Hypertonic saline will be non-inferior to mannitol in decreasing elevated ICP.

Secondary hypotheses:

1. Hypertonic saline therapy will result with fewer complications than mannitol
2. ICP reduction duration will be longer using hypertonic saline when compared with mannitol

DETAILED DESCRIPTION:
There is growing evidence in the literature indicating that ICP and Cerebral Perfusion Pressure measurements may not be sufficient in the management of elevated ICP. Based on this evidence, monitoring of partial brain tissue oxygenation has gain acceptance among neurosurgeons and neurointensivists, and has become a standard of care monitor in some centers across the country. There is, however, insufficient information in the literature describing the effects of hyperosmolar medications on regional brain tissue oxygenation.

We intend to undertake this non-inferiority, prospective, randomized double-blind study to answer very important clinical questions not yet answered in the literature: Will hypertonic saline therapy, given at equiosmolar load, be non-inferior to mannitol in reducing elevated ICP?

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* elevated ICP requiring ICP monitoring
* ICP ≥ 25 mmHg 5 min after ICP bolt or EVD placement

Exclusion Criteria:

* Requiring decompressive craniotomy or post decompressive craniotomy
* Hyponatremia (sodium level < 125 mEq/L)
* Hypernatremia (sodium > 155 mmol/L)
* Serum osmolality ≤ 250 mOsm/kg
* Serum osmolality ≥ 320 mOsm/kg
* Physical exam compatible with brain death
* Patients on hemodialysis with end-stage renal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Percent reduction of ICP from baseline | 30 minutes from completion of medication administration

SECONDARY OUTCOMES:
Time from study drug administration completion to ICP < 25 mmHg | First 72 hours
Cumulative duration of ICP below 25 mmHg | First 24 hours
Cumulative duration of ICP below 25 mmHg | First 72 hours
Cumulative duration of cerebral perfusion pressure (CPP) above 60 mmHg | First 24 hours
Cumulative duration of cerebral perfusion pressure (CPP) above 60 mmHg | First 72 hours
Cumulative duration of regional oxygen partial pressure (pbtO2) > 20% | two hours following each dose administration during the first 24 hours
Total dose of medications given | First 24 hours; also over 3 days
Frequency of treatment failure | First 72 hours
  Treatment failure defined as ICP > 30 mmHg for > 30 minutes
Frequency of rebound intracranial hypertension | First 72 hours
  Rebound intracranial hypertension defined as ICP > 25 mmHg for more than 10 minutes following ICP stabilization
Frequency of composite Major Adverse Events | 3 days
  1. acute kidney injury as defined by an increase in creatinine x 2 or GFR decrease > 50% or urine output < 0.5 ml/kg/h for 12 hours, compared to baseline, as per RIFLE criteria
  2. hypotensive episodes (SBP < 90 mmHg for more than 10 minutes)
  3. hemodynamic instability as measured by decrease of cardiac output by more than 15% within two hours following medication administration
  4. pulmonary edema as defined by ELWI I> 10
Difference in inflammatory response | Regular intervals over first 3 days
  Determined by analysis of cytokine and inflammatory biomarkers.
Difference in average pre-discharge stroke scale score | hospital discharge (or 30 days if not discharged)

CONTACTS AND LOCATIONS:
Overall Officials: Achikam Oren-Grinberg, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shackford SR, Bourguignon PR, Wald SL, Rogers FB, Osler TM, Clark DE. Hypertonic saline resuscitation of patients with head injury: a prospective, randomized clinical trial. J Trauma. 1998 Jan;44(1):50-8. doi: 10.1097/00005373-199801000-00004. PMID 9464749
- [Background] BARRY KG, BERMAN AR. Mannitol infusion. III. The acute effect of the intravenous infusion of mannitol on blood and plasma volumes. N Engl J Med. 1961 May 25;264:1085-8. doi: 10.1056/NEJM196105252642105. No abstract available. PMID 13687351
- [Background] Brain Trauma Foundation; American Association of Neurological Surgeons; Congress of Neurological Surgeons; Joint Section on Neurotrauma and Critical Care, AANS/CNS; Bratton SL, Chestnut RM, Ghajar J, McConnell Hammond FF, Harris OA, Hartl R, Manley GT, Nemecek A, Newell DW, Rosenthal G, Schouten J, Shutter L, Timmons SD, Ullman JS, Videtta W, Wilberger JE, Wright DW. Guidelines for the management of severe traumatic brain injury. II. Hyperosmolar therapy. J Neurotrauma. 2007;24 Suppl 1:S14-20. doi: 10.1089/neu.2007.9994. No abstract available. PMID 17511539
- [Background] The Brain Trauma Foundation. The American Association of Neurological Surgeons. The Joint Section on Neurotrauma and Critical Care. Use of mannitol. J Neurotrauma. 2000 Jun-Jul;17(6-7):521-5. doi: 10.1089/neu.2000.17.521. PMID 10937895
- [Background] Bereczki D, Liu M, Prado GF, Fekete I. Cochrane report: A systematic review of mannitol therapy for acute ischemic stroke and cerebral parenchymal hemorrhage. Stroke. 2000 Nov;31(11):2719-22. doi: 10.1161/01.str.31.11.2719. PMID 11062300
- [Background] Qureshi AI, Suarez JI, Bhardwaj A, Mirski M, Schnitzer MS, Hanley DF, Ulatowski JA. Use of hypertonic (3%) saline/acetate infusion in the treatment of cerebral edema: Effect on intracranial pressure and lateral displacement of the brain. Crit Care Med. 1998 Mar;26(3):440-6. doi: 10.1097/00003246-199803000-00011. PMID 9504569
- [Background] Huang SJ, Chang L, Han YY, Lee YC, Tu YK. Efficacy and safety of hypertonic saline solutions in the treatment of severe head injury. Surg Neurol. 2006 Jun;65(6):539-46; discussion 546. doi: 10.1016/j.surneu.2005.11.019. PMID 16720165